CLINICAL TRIAL: NCT07086638
Title: ROS-Scavenging Nanozyme Combined With Near-Infrared Thermotherapy for the Amelioration of Grade III Radiation Dermatitis in Patients With Head and Neck Cancer
Brief Title: ROS-Scavenging Nanozyme Combined With Thermotherapy Alleviate Radiation Dermatitis in Patients With Head and Neck Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-134-2
Record Dates: First submitted 2025-07-15; First posted 2025-07-25 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-07

CONDITIONS: Radiation Dermatitis
MeSH Terms: conditions — Radiodermatitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Photo-responsive nanozyme (Experimental): The nanozyme scavenges ROS at the site of dermatitis and simultaneously responds to NIR light to generate mild heat, thereby promoting the healing of radiation-induced skin injury.
  Interventions: Drug: Photo-responsive nanozyme

INTERVENTIONS:
Drug: Photo-responsive nanozyme — The nanozyme scavenges ROS at the site of dermatitis and simultaneously responds to NIR light to generate mild heat, thereby promoting the healing of radiation-induced skin injury.

SUMMARY:
Severe radiation dermatitis remains a challenging complication in head and neck cancer with limited treatment options; this study aims to evaluate a novel Prussian blue-based nanozyme combined with near-infrared thermotherapy to promote effective healing of Grade III lesions.

DETAILED DESCRIPTION:
Radiation dermatitis is a common and challenging complication for patients undergoing radiotherapy, especially those with head and neck cancer. Currently, there are limited effective clinical treatments available for managing severe (Grade III) radiation-induced skin damage.

This study aims to explore a novel and safe treatment strategy for alleviating Grade III radiation dermatitis. The investigators use Prussian blue, an FDA-approved compound known for its reactive oxygen species (ROS) scavenging ability, formulated into a nanozyme that targets oxidative stress at the injury site. When combined with near-infrared (NIR) thermotherapy, this approach promotes faster skin repair and reduces inflammation.

This study's goal is to provide an effective and patient-friendly therapeutic option that accelerates healing and improves quality of life for individuals suffering from severe radiation dermatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a pathological diagnosis of non-metastatic head and neck malignant tumors;
2. Patients deemed suitable for high-dose radiotherapy, either as a primary treatment or as postoperative treatment following surgical resection.

Exclusion Criteria:

1. Eastern Cooperative Oncology Group performance status of >2;
2. Pre-existing skin rash, ulceration or open wound in the treatment area;
3. Known allergy to trolamine or prussian blue;
4. Inflammatory or connective tissue disorder of the skin;
5. History of head and neck radiotherapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2025-09-25 (Estimated); Study Completion 2025-10-25 (Estimated)

PRIMARY OUTCOMES:
The incidence of grade 3 radiation dermatitis | From the onset of Grade III dermatitis to two weeks after the completion of radiotherapy
  Patients are assessed weekly for radiation dermatitis by an experienced radiation oncology nurse according to the Radiation Therapy Oncology Group (RTOG) criteria.

SECONDARY OUTCOMES:
Bacterial load at the site of dermatitis | From the first administration of drug treatment through study completion, an average of 1 month.
  Experienced radiation oncology nurses took samples from the patients' radiation dermatitis areas, and professional medical laboratory nurses performed bacterial load analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Xingchen Peng, Principal Investigator — Sichuan University West China Hospital
Locations (1):
- Sichuan University West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No